CLINICAL TRIAL: NCT06589362
Title: Enhancing Cognitive Rehabilitation After TBI Using Noninvasive Vagal Nerve Stimulation
Brief Title: Noninvasive Vagal Nerve Stimulation and Cognitive Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Shira Cohen-Zimerman, Research Scientist, PhD, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU00221084
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: a single-blind sham-controlled randomized crossover pilot study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transcutaneous auricular vagus nerve stimulation (Active Comparator): Active vagus nerve stimulation.
  Interventions: Device: Transcutaneous auricular vagus active nerve stimulation
- Sham Transcutaneous auricular vagus nerve stimulation (Sham Comparator): Sham vagus nerve stimulation.
  Interventions: Device: Transcutaneous auricular vagus sham nerve stimulation

INTERVENTIONS:
Device: Transcutaneous auricular vagus active nerve stimulation — In the active stimulation, two electrodes are placed in the cymba conchae of one of the ears, an area thought to be exclusively innervated by the auricular branch of the vagus nerve.
  Arms: Transcutaneous auricular vagus nerve stimulation
Device: Transcutaneous auricular vagus sham nerve stimulation — In the sham stimulation, the electrodes are placed on the tail of helix, which is free of vagal innervation.
  Arms: Sham Transcutaneous auricular vagus nerve stimulation

SUMMARY:
The purpose of this study is to examine the feasibility and preliminary efficacy of using transcutaneous auricular vagus nerve stimulation (tVNS) to enhance cognitive recovery in patients with mild-moderate traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Eligible participants will be invited to two sessions, 2-7 days apart. In each session, either active tVNS or sham stimulation will be administered while the participants are performing tasks of executive functions. The order of the sessions (tVNS vs Sham) will be counterbalanced across participants.

ELIGIBILITY:
Inclusion Criteria:

In inpatient rehabilitation due to recent Traumatic Brain Injury, ages 18-65 years.

Ability to independently use a keyboard. Able to understand and communicate in English (according to clinical judgment). Able to independently provide consent to participate. Orientation to place, time, and situation (two consecutive scores of 25 or more on the Orientation Log(O-Log)40. This scale is routinely administered during acute rehabilitation stay.

Exclusion criteria:

Acute medical issues requiring close physician or nursing monitoring. Bioelectrical implants, including pacemakers. Pregnancy or persons who are lactating. Significant gross or fine motor weakness. Significant, ongoing communication or comprehension impairments (such as aphasia) that would affect an individual's ability to complete the required assessments.

Acute agitation or behavioral issues, as defined by a last Agitated Behavior Scale Score greater than 21 (routinely administered during acute rehabilitation stay, that would affect an individual's ability to participate in the required assessments.

Severely impaired memory retention (Score lower than 3 in the 3 Word Delayed Recall test, routinely administered during acute rehabilitation stay.

Diagnosis of depression. Active substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
N-Back Computerized Task | 15 minutes
  In the n-back task, participants are presented a series of visual stimuli. They are asked for each stimulus whether it matches a stimulus n trials before. For example, in a 2-back task, in which the trials consist of letters, participants have to decide whether the current letter is the same as the letter in trial n - 2. We will use a computerized version of this task.
Trail Making Test - Parts A & B | 5 minutes
  Trail Making Part A requires participants to draw a line between circles containing numbers in ascending order (e.g., 1-2- 3...etc.). Part B requires participants to alternate drawing a line between ascending letters and numbers (e.g., 1-A-2-B...etc.). The key measures are the time required to complete and the number of errors made in Part A and Part B. This test measures various aspects of cognition including attention, visual search, motor coordination, reasoning, and task-switching.

CONTACTS AND LOCATIONS:
Overall Officials: Shira Cohen-Zimerman, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States